CLINICAL TRIAL: NCT00793728
Title: Prospective Randomized Trial Comparing Two Techniques of Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Amador Garci-a Ruiz de Gordejuela, MD, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR131/08
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Morbid Obesity
Keywords: Morbid obesity; High risk
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antrectomy (Active Comparator)
  Interventions: Procedure: Sleeve gastrectomy
- Without antrectomy (Active Comparator)
  Interventions: Procedure: Sleeve gastrectomy

INTERVENTIONS:
Procedure: Sleeve gastrectomy — Perform a gastrectomy guided by a 38F catheter and parallel to the small curvature of the stomach

SUMMARY:
This study compares if there is any difference doing antrectomy while performing a sleeve gastrectomy for treating morbid obesity. The investigators compare the differences between leaving or not leaving the antrum in terms of food tolerance, weight lost and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* BMI>40 kg/m2
* Age >18 years old
* Eligible for laparoscopic surgery

Exclusion Criteria:

* Prior bariatric surgery
* Sleeve gastrectomy as a part of a duodenal switch
* Second time surgery before 18 months
* Other procedures done during the surgery
* Conversion to laparotomy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2008-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Weight lose | One year
Food tolerance | One year
Quality of life | One year

SECONDARY OUTCOMES:
Metabolic syndrome outcome | One year

CONTACTS AND LOCATIONS:
Overall Officials: Amador Garcia Ruiz de Gordejuela, Consultant, Principal Investigator — Consultant of Surgery; Jordi Pujol Gebelli, Consultant, Principal Investigator — Consultant of Surgery; Carles Masdevall Noguera, Consultant, Principal Investigator — Consultant of Surgery
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain